CLINICAL TRIAL: NCT01487070
Title: A Single-Center Trial of Intravitreous Injections of Macugen (Pegaptanib Sodium) Given at Least 7 Days Before Vitrectomy Secondary To Tractional Retinal Detachment in Proliferative Diabetic Retinopathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Retina Institute of Hawaii (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIH1005
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-04

CONDITIONS: PDR
MeSH Terms: interventions — pegaptanib

ARMS (1):
- Macugen (Pegaptanib Sodium) (Experimental): Open-label, single-center trial. Subjects will recieve intravitreous injections of Macugen 7-14 days before Vitrectomy.
  Interventions: Drug: Macugen (Pegaptanib Sodium)

INTERVENTIONS:
Drug: Macugen (Pegaptanib Sodium) — Pegaptanib sodium drug substance is a pegylated (40 kDa branched PEG molecule consisting of two 20 kDa PEG arms) anti-VEGF aptamer. It is formulated in phosphate buffered saline at pH 6-7. Sodium hydroxide or hydrochloric acid may be added for pH adjustment.
  Pegaptanib sodium is formulated at 0.3mg/90µl and presented in a USP Type I glass barrel syringe sealed with a bromobutyl rubber stopper. A 30-guage needle is fixed to the end of the syringe after removal of the rubber stopper. The syringe comes in a sealed foil pouch, and the 30-gauge needle is added to the sterile injection field separately. The drug product is preservative-free and intended for single use by intravitreous injection only.

SUMMARY:
Primary objective of this trial will be to evaluate the safety and efficacy of intravitreal injections of Macugen (pegaptanib sodium) when given at least 7-14 days prior to vitrectomy in subjects with tractional retinal detachment (with or withoutmacular involvement) secondary to proliferative diabetic retinopathy.

Secondary objective is to evaluate regression of neovascularization and progression of macular traction utilizing OCT and fundus photographs.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either gender aged 75 years or below diagnosed with tractional retinal detachment secondary to proliferative diabetic retinopathy.

Exclusion Criteria:

* Subjects with vitreous hemorrhage obscuring the posterior pole will be excluded.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Evidence of advancement of tractional detachment post injection of Macugen before surgical intervention. | 7-14 days prior to surgical intervention

SECONDARY OUTCOMES:
Evaluate regression of neovascularization and progression of macular traction utilizing OCT and Fundus photographs | 7-14 days prior to surgical intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Retina Institute of Hawaii, Honolulu, Hawaii, United States